CLINICAL TRIAL: NCT07111377
Title: The Efficacy of Brief Cognitive Behavioral Therapy (Brief CBT) in Reducing Suicidal Ideation Among Economically Distressed Migrant Workers in the Middle East: A Randomized Controlled Trial
Brief Title: Brief Cognitive Behavioral Therapy for Reducing Suicidal Ideation in Economically Distressed Migrants
Acronym: Brief CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bath Spa University Academic Centre RAK (Other)
Responsible Party: Principal Investigator, Jamal D. Magantor, Program Leader , Department of Psychology, Bath Spa, Bath Spa University Academic Centre RAK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSU-RAK-PSYCH - 2025-0008
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Suicidal Ideation; Depression; Anxiety; Financial Stress
Keywords: Suicidal Ideation; Migrant Workers; Brief Cognitive Behavioral Therapy; Financial Stress
MeSH Terms: conditions — Suicidal Ideation; Depression; Anxiety Disorders; Financial Stress

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned (1:1) to either Brief CBT or Treatment as Usual (TAU).
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors were blinded to group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief CBT (Experimental): Participants assigned to this arm received an 8-session culturally adapted Brief Cognitive Behavioral Therapy (Brief CBT). Sessions addressed crisis stabilization, cognitive restructuring, problem-solving related to financial stressors, behavioral activation, emotion regulation skills, relapse prevention, and linkage to community resources. Sessions were delivered weekly, either individually (60 minutes) or in groups (90 minutes), based on participant preference.
  Interventions: Behavioral: Brief Cognitive Behavioral Therapy
- Treatment as Usual (TAU) (No Intervention): Participants assigned to this arm received standard community resources and information without structured therapeutic intervention. They were provided with a comprehensive multilingual list of available mental health services, crisis support hotlines, and financial counseling resources accessible in the UAE. Participants were free to access these services independently, without active facilitation or structured guidance by the research team. This arm represents the standard of care typically available to economically distressed migrant workers experiencing mental health difficulties in the region.

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Therapy — Participants received an 8-session culturally adapted Brief Cognitive Behavioral Therapy intervention targeting suicidal ideation, psychological distress, and financial stress. Therapy included crisis stabilization, cognitive restructuring of maladaptive thoughts related to economic hardship, behavioral activation, problem-solving skills for financial and psychosocial stressors, and emotion-regulation training. It concluded with relapse prevention planning and connection to supportive community resources. Sessions were delivered weekly, either individually (60 minutes) or in groups (90 minutes), based on participant preference.
  Arms: Brief CBT

SUMMARY:
This randomized controlled trial assessed the efficacy of an 8-session, culturally adapted Brief Cognitive Behavioral Therapy (Brief CBT) compared to Treatment as Usual (TAU) in reducing suicidal ideation among economically distressed migrant workers in the United Arab Emirates. Participants (N=120) were randomized to receive Brief CBT or TAU. Outcomes were assessed at baseline, 4-weeks, 8-weeks, and 3-month follow-up.

DETAILED DESCRIPTION:
Economically distressed migrant workers face high psychosocial stress, resulting in increased suicidal ideation. This study examined the effectiveness of culturally adapted Brief CBT in addressing suicidal ideation, depression, anxiety, stress, and financial distress compared to standard treatment resources provided as usual.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 65 years.
* Migrant worker residing in the UAE with a valid work or residence visa.
* Experiencing significant economic distress (score of ≤40 on the InCharge Financial Distress/Financial Well-Being Scale - IFDFW).
* Presence of suicidal ideation, defined as a score ≥1 on the Beck Scale for Suicide Ideation (BSS).
* Able to communicate effectively in English, Arabic, or Tagalog.
* Willing and able to provide informed written consent.

Exclusion Criteria:

* Acute psychosis, severe substance dependence, or immediate suicide risk requiring hospitalization.
* Cognitive impairment limiting therapy participation.
* Currently engaged in structured psychotherapy for depression or suicidality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Reduction in Suicidal Ideation Severity (Beck Scale for Suicide Ideation; BSS) | Baseline, 4 weeks (mid-treatment), 8 weeks (post-treatment), and 3-month follow-up
  Change in the severity of suicidal ideation as measured by the Beck Scale for Suicide Ideation (BSS), a 19-item clinician-rated scale that assesses suicidal thoughts, plans, and wishes during the past week. Scores range from 0 to 38, with higher scores indicating greater suicidal ideation severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Bath Spa University Academic Centre RAK, Dubai, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bryan CJ, Rudd MD. Brief Cognitive-Behavioral Therapy for Suicide Prevention. New York: The Guilford Press; 2018.
- [Background] Prawitz AD, Garman ET, Sorhaindo B, O'Neill B, Kim J, Drentea P. InCharge Financial Distress/Financial Well-Being Scale: Development, administration, and score interpretation. Journal of Financial Counseling and Planning. 2006;17(1):34-50.
- [Background] Lovibond SH, Lovibond PF. Manual for the Depression Anxiety Stress Scales. 2nd ed. Sydney: Psychology Foundation; 1995.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Beck AT, Steer RA, Ranieri WF. Scale for Suicide Ideation: psychometric properties of a self-report version. J Clin Psychol. 1988 Jul;44(4):499-505. doi: 10.1002/1097-4679(198807)44:43.0.co;2-6. PMID 3170753